CLINICAL TRIAL: NCT01926119
Title: TMS for CRPS - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Chief, Division of Pain Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25894
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Complex Regional Pain Syndrome (CRPS)
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Transcranial Magnetic Stimulation

ARMS (1):
- TMS Intervention - 5 days (Experimental): Application of Transcranial Magnetic Stimulation (TMS) once per day over 5 days.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation

SUMMARY:
The purpose of this pilot study is to test whether Transcranial Magnetic Stimulation (TMS) may alleviate the symptoms of Complex Regional Pain Syndrome (CRPS). The investigators will test various methods of TMS in a small pilot study to investigate what methods may have clinical potential. This is a small pilot study to determine feasibility and signal to potentially inform future trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Diagnosis of CRPS (complex regional pain syndrome)
3. Average pain level reported on Numerical Rating Scale meets entry criteria
4. Ability to perform the experimental task and procedures.

Exclusion Criteria:

1. MRI contraindication (metal implants or devices, claustrophobia)
2. TMS Contraindication (eg metal implant or devices near the site of stimulation)
3. History of epilepsy
4. History of a psychological or psychiatric disorder that would interfere with study procedures, at the discretion of the researcher.
5. Neurologic illness that would interfere with brain integrity
6. Current medical condition or medication use that would interfere with study procedures or data integrity, at the discretion of the researcher.
7. Currently pregnant or planning to become pregnant.
8. On going legal action or disability claim.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS Intervention - 5 Days: Application of Transcranial Magnetic Stimulation (TMS) once per day over 5 days in the order of Theta Burst Stimulation followed by High frequency stimulation
  Transcranial Magnetic Stimulation
Period: Overall Study
Arm/Group | TMS Intervention - 5 Days
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TMS Intervention - 5 Days
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 55.5 [48 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain
Description: Numerical rating scale (NRS) where 0=no pain and 10=worst pain imaginable
Time Frame: Baseline to post-TMS day 5
Population: Completed 5 days of TMS
Measure: Mean (Full Range); unit: units on a scale
Groups:
- TMS Intervention - 5 Days: Application of Transcranial Magnetic Stimulation (TMS) once per day over 5 days.
  Transcranial Magnetic Stimulation
Arm/Group | TMS Intervention - 5 Days
Number analyzed (Participants) | 3
units on a scale
  Baseline NRS | 5.2 [3.6 to 7.2]
  Post-TMS day 5 NRS | 0.7 [0 to 1.1]

2. Secondary Outcome: Change in Motor Function and Coordination
Description: As assessed by functional capacity exam and physical exam
Time Frame: End of 5-day treatment series and at 1-week follow-up relative to baseline
Population: This data was not collected and was therefore not analyzed.
Arm/Group | TMS Intervention - 5 Days
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Sensory Perception
Time Frame: End of each treatment session and at 1-week follow-up as compared to baseline
Population: This data was not collected and therefore not analyzed.
Arm/Group | TMS Intervention - 5 Days
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Vasomotor Function
Time Frame: End of each treatment session and at 1-week follow-up as compared to baseline
Population: This data was not collected and therefore not analyzed.
Arm/Group | TMS Intervention - 5 Days
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Sudomotor Function
Time Frame: End of each treatment session and at 1-week follow-up as compared to baseline
Population: This data was not collected and therefore not analyzed.
Arm/Group | TMS Intervention - 5 Days
Number analyzed (Participants) | 0

6. Secondary Outcome: Trophic Changes
Time Frame: End of each treatment session and at 1-week follow-up as compared to baseline
Population: This data was not collected and therefore not analyzed.
Arm/Group | TMS Intervention - 5 Days
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Motor Strength and Joint Range of Motion
Time Frame: End of each of the 5 treatment sessions and at 1-week follow-up relative to baseline
Population: This data was not collected and therefore not analyzed.
Arm/Group | TMS Intervention - 5 Days
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants were followed during 5 days of treatment and for 1 week following treatment
Description: Participants were assessed for pain before and after each treatment session and at 1 week follow-up. During these assessments adverse events were evaluated as well.
Arm/Group | TMS Intervention - 5 Days
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS Intervention - 5 Days (N=4)
Headache (Nervous system disorders) | 3 (3) — participants reported headache after stimulation
Nausea and vomiting (Gastrointestinal disorders) | 2 (2) — participants reported nausea and vomiting 6-8 hours after treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes